CLINICAL TRIAL: NCT06506591
Title: A Single-And Multiple-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics,Pharmacodynamics and Food Effect of WD-890 Tablets in Healthy Chinese Subjects
Brief Title: A Single-And Multiple-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Food Effect of WD-890 Tablets in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang Wenda Pharma Technology LTD. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: WENDA890ZQ
Record Dates: First submitted 2024-06-28; First posted 2024-07-17 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Healthy Participants
Keywords: TYK2 Inhibitor

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: SAD and MAD ：Double (Participant,Investigator) FE：Open Label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- WD-890 1mg (Experimental): Take a fixed dose of WD-890 tablets orally
  Interventions: Drug: WD-890
- WD-890 3mg (Experimental): Take a fixed dose of WD-890 tablets orally
  Interventions: Drug: WD-890
- WD-890 6mg (Experimental): Take a fixed dose of WD-890 tablets orally
  Interventions: Drug: WD-890
- WD-890 9mg (Experimental): Take a fixed dose of WD-890 tablets orally
  Interventions: Drug: WD-890
- WD-890 Tablets Placebo (Placebo Comparator): Take a fixed dose of WD-890 tablets Placebo orally
  Interventions: Drug: WD-890 Tablets Placebo

INTERVENTIONS:
Drug: WD-890 — Administered P.O.
  Arms: WD-890 1mg; WD-890 3mg; WD-890 6mg; WD-890 9mg
Drug: WD-890 Tablets Placebo — Administered P.O.
  Arms: WD-890 Tablets Placebo

SUMMARY:
This is a phase I, randomised, double-blind, placebo-controlled, 3-part study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics and food effect of WD-890 Tablets in Healthy Chinese Subjects

ELIGIBILITY:
Inclusion Criteria：

* Signed Informed Consent.
* 18 Years to 50 Years (Adult).
* Body mass index (BMI) of 19 to 26 kg/m2, inclusive, and total body weight ：male >=50 kg; female >= 45.0 kg.

Exclusion Criteria：

* Has any surgery performed within 6 months prior to screening, or during the study period.
* Inability to swallow solid tablets.
* Inability to be venipunctured and tolerate venous access.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2023-10-26 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Safety of a single oral dose of WD-890 based on number of incidence of AE, SAEs, marked abnormalities in clinical laboratory tests, vital sign measurements, ECGs, telemetry, and physical examinations | Days 1 to 5
Tolerability of a single oral dose of WD-890 based on number of incidence of AE, SAEs, marked abnormalities in clinical laboratory tests, vital sign measurements, ECGs, telemetry, and physical examinations | Days 1 to 5
Safety of a multiple oral dose of WD-890 based on number of incidence of AE, SAEs, marked abnormalities in clinical laboratory tests, vital sign measurements, ECGs, telemetry, and physical examinations | Days 1 to 19
Tolerability of a multiple oral dose of WD-890 based on number of incidence of AE, SAEs, marked abnormalities in clinical laboratory tests, vital sign measurements, ECGs, telemetry, and physical examinations | Days 1 to 19
Single Ascending Dose (SAD), Multiple Ascending Dose (MAD) and Food Effect (FE) Cohorts: Maximum Observed Plasma Concentration (Cmax) of WD-890； | SAD: Days 1 to 4 ; MAD: Day 1, Day 6, Day 9 and Day 12; FE: Days 1 to 5, Days 8 to 12
Single Ascending Dose (SAD), Multiple Ascending Dose (MAD) and Food Effect (FE) Cohorts: Area Under The Plasma Concentration-Time Curve From Time Zero to Time of Last Quantifiable Concentration (AUC(0-T)) of WD-890 | SAD: Days 1 to 4 ; MAD: Day 1, Day 6, Day 9 and Day 12 FE: Days 1 to 5, Days 8 to 12
Single Ascending Dose (SAD), Multiple Ascending Dose (MAD) and Food Effect (FE) Cohorts: Area Under The Plasma Concentration-Time Curve From Time Zero Extrapolated To Infinite Time (AUC(INF)) of WD-890 | SAD: Days 1 to 4 ; MAD: Day 1, Day 6, Day 9 and Day 12 FE: Days 1 to 5, Days 8 to 12
Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) Cohorts: Time to Maximum Observed Plasma Concentration (Tmax) of WD-890 | SAD: Days 1 to 4 ; MAD: Day 1, Day 6, Day 9 and Day 12
Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) Cohorts: Apparent Plasma Elimination Half-Life (T-HALF) of WD-890 | SAD: Days 1 to 4 ; MAD: Day 1, Day 6, Day 9 and Day 12
Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) Cohorts: Apparent Volume of Distribution (Vz/F) of WD-890 | SAD: Days 1 to 4 ; MAD: Day 1, Day 6, Day 9 and Day 12
Multiple Ascending Dose (MAD) Cohorts: Maximum Observed Plasma Concentration at Steady State (Cmax,ss) of WD-890 | Day 1, Day 6, Day 9 and Day 12
Multiple Ascending Dose (MAD) Cohorts: Time to Reach the Maximum Plasma Concentration at Steady State (Tmax,ss) of WD-890 | Day 1, Day 6, Day 9 and Day 12
Multiple Ascending Dose (MAD) Cohorts: Apparent Volume of Distribution at Steady State (Vss/F) of WD-890 | Day 1, Day 6, Day 9 and Day 12

SECONDARY OUTCOMES:
Food Effect Cohorts: Time to Maximum Observed Plasma Concentration (Tmax) of WD-890 | Days 1 to 5, Days 8 to 12,
Food Effect Cohorts: Apparent Volume of Distribution (Vz/F) of WD-890 | Days 1 to 5, Days 8 to 12
Food Effect Cohorts: Apparent Plasma Elimination Half-Life (T-HALF) of WD-890 | Days 1 to 5, Days 8 to 12,

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No